CLINICAL TRIAL: NCT00685724
Title: A Pilot SMART Design for Pathological Gamblers
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 07-259; P50DA009241 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Pathological Gambling
Keywords: pathological gambling; cognitive-behavioral therapy; motivational enhancement therapy
MeSH Terms: conditions — Gambling | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Following 2 sessions of MET intervention received by all patients, patients in Condition 1 receive no further intervention.
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)
- 2 (Experimental): Patients in Condition 2 will receive 8 sessions of the CBT (Cognitive Behavioral Therapy) intervention.
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)
- 3 (Experimental): Patients in Condition 3 will receive 8 sessions of CBT plus aftercare treatment.
  Interventions: Behavioral: Motivational Enhancement Therapy (MET); Behavioral: Cognitive-Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy (MET) — MET is a client-centered, directive form of therapy designed to enhance clients' intrinsic motivation to change.
Behavioral: Cognitive-Behavioral Therapy (CBT) — In CBT, clients learn to modify their thoughts as well as their behaviors by increasing awareness of the relationship between thoughts, emotions, and actions.
  Arms: 3

SUMMARY:
Pathological gambling is serious problem, with significant psychological, financial, and public health consequences. Nevertheless, controlled trials examining the efficacy of therapeutic interventions for pathological gamblers are sparse, and many pathological gamblers recover on their own, or with only minimal interventions. In this initial study of a SMART design for pathological gamblers, we will offer a brief intervention to all (n = 100), and subsequently randomize individuals based upon their initial treatment response to varying intensities of additional care from none to 8 sessions of individual cognitive behavioral therapy (CBT) plus 14 weeks of Aftercare. Gambling outcomes will be assessed pre-treatment and at about weeks 10, 24, 36 and 52.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old, DSM-IV criteria for pathological gambling
* >2 gambling episodes in past 60 days
* spent >$100 wagering in the past 60 days
* willingness to accept random assignment after the brief intervention.

Exclusion Criteria:

* Reading level below 5th grade
* uncontrolled psychiatric conditions (e.g., active suicidal intention, psychosis, bipolar disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
self and collateral indices of gambling and gambling related problems | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States